CLINICAL TRIAL: NCT02662842
Title: BD FlowSmart™ User Claims Study
Brief Title: BD FlowSmart™ Subcutaneous Insulin Infusion Set User Preference and Claims Study
Status: Completed | Type: Observational
Sponsor: Becton, Dickinson and Company (Industry)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Other Study IDs: DBC-15SCARL15
Record Dates: First submitted 2016-01-19; First posted 2016-01-26 (Estimated); Last update posted 2017-04-13 (Actual); Status verified 2017-04

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: infusion set; continuous subcutaneous insulin infusion
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- FlowSmart Infusion set, then current set: Subjects will use the FlowSmart Infusion Set for a period of 9 to 11 days, then switch to their current infusion set for another period of 9 to 11 days. Subjects must use at least 3 sets during each Study Period then - Subjects will use their current infusion set for a period of 9 to 11 days, then switch to the FlowSmart infusion set for another period of 9 to 11 days. Subjects must use at least 3 sets during each Study Period.
  Interventions: Device: FlowSmart Infusion Set; Device: Current Infusion Set

INTERVENTIONS:
Device: FlowSmart Infusion Set — Use of set for subcutaneous insulin infusion, with set change every three days.
Device: Current Infusion Set — Use of set for subcutaneous insulin infusion, with set change every three days.

SUMMARY:
Continuous Subcutaneous Insulin Infusion (CSII) via insulin pump therapy has been shown to improve quality of life and glucose control in many patients with diabetes opting for this treatment modality. Despite significant innovation and advancement in pump technology, insulin infusion sets have been an area where innovation has been significantly lacking with no clinical studies performed prior to product launches.

BD has developed a subcutaneous infusion set with FlowSmart™ Technology designed to address patient comfort, insulin delivery and flow interruptions. According to preliminary animal and clinical studies, this technology results in lower infusion pressure indicating more consistent insulin delivery.

The FlowSmart infusion set has been previously tested in prototype form with healthy non-diabetic subjects with the sets inserted by nurses, and with CSII-using patients who self-inserted the FlowSmart infusion set in a clinical research setting.

The purpose of this study is to determine if insulin pump users prefer using the BD FlowSmart infusion set compared to their current set with respect to insertion pain and wear comfort.

ELIGIBILITY:
Inclusion Criteria:

* Must be 18-75 years of age, inclusive
* Have type 1 diabetes
* Treating diabetes with CSII for at least 12 months
* Currently using a soft catheter infusion set that is inserted 90° to body surface
* Have HbA1c ≤ 9.0% (tested at enrollment)
* Willing to do self monitoring of blood glucose (SMBG) using the supplied BG meter
* Able to read, write and follow instructions in English
* Able and willing to provide informed consent
* Willing to use each infusion set (both study and current) for 72 hours (3 days)
* Willing to use their usual insertion method (manual or mechanical inserter) with both infusion sets

Exclusion Criteria:

* Pregnant (pre-menopausal females only; tested at enrollment)
* Recent history (within 6 months) of unstable diabetes including ketoacidosis, hyperglycemia and/or hypoglycemia requiring hospitalization(self-reported)
* Physical conditions that restrict dexterity and may limit ability to perform study procedure (e.g., severe neuropathy or arthritis of the hands, self-reported)
* Any other condition the PI or designee deems to pose a risk to the subject in the study
* Currently taking steroidal medications (self-reported)
* Acutely ill as determined by the Principal Investigator.
* Currently using an insulin infusion pump whose insulin reservoir is not compatible with either a Paradigm or Luer connector, such as Sooil Dana, Asante Snap, and Accu-Chek insight
* Currently using a disposable (patch) insulin pump, such as the Insulet Omnipod and the Valeritas V-Go
* Currently using a Teflon infusion set that is not inserted at a 90° angle, such as the Animas Comfort, Animas Inset 30, Medtronic Silhouette, or a steel infusion set, such as the Accu-Chek Rapid-D or Medtronic Sure-T
* Currently using Advanced Diabetes Research (ADR) reservoirs
* Currently participating in any other clinical investigations that conflicts with this one, or who have participated in a study with the same indication within the last 3 months and that the Principal Investigator or designee believes will conflict with outcomes or ability of the subject to complete all activities required in the study
* Participated in one or more of the following BD studies: DBC-14SCARL10 and DBC-14SCARL13
* Employed by, or currently serving as a contractor or consultant to BD or study site

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 75 subjects with type 1 diabetes currently on CSII will participate in the study
Enrollment: 75 (Actual)
Dates: Start 2016-01; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Comparative Infusion Set Insertion Pain | Comparative pain measure assessed at the end of Study Period 2, after 9-11 days use of each infusion set type
  At the study visit after completing both study periods (Visit 3), subjects will use a 15 cm Visual Analog Scale (VAS) to indicate which insertion set was less painful to insert, the BD Flowsmart or their current infusion set. Effects of infusion set type will be tested for statistical significance using linear mixed models adjusting for the effect of subject, study site and period. The model will be used to generate a two-sided 95% confidence interval for the adjusted average pain rating using a multiple comparison approach.
Comparative Infusion Set Wear Comfort | Comparative pain measure assessed at the end of Study Period 2, after 9-11 days use of each infusion set type
  At the study visit after completing both study periods (Visit 3), subjects will use a 15 cm Visual Analog Scale (VAS) to indicate which set was more comfortable to wear, the BD FlowSmart or their current infusion set. Only if reduced Pain (outcome 1) for FlowSmart if achieved will wear comfort be further analyzed. Effects of infusion set type will be tested for statistical significance using linear mixed models adjusting for the effect of subject, study site and period. The model will be used to generate a two-sided 95% confidence interval for the adjusted average comfort rating using a multiple comparison approach.

SECONDARY OUTCOMES:
Overall Infusion Set Preference | Assessed at the end of Study Period 2, after 9-11 days use of each infusion set type
  At the study visit after completing both study periods (Visit 3), subjects will use a 15 cm Visual Analog Scale (VAS) to indicate their preference for the BD Flowsmart compared to their current infusion set based on their recent experience. Effects of infusion set type will be tested for statistical significance using linear mixed models adjusting for the effect of subject, study site and period. The model will be used to generate a two-sided 95% confidence interval for the adjusted preference rating using a multiple comparison approach.

CONTACTS AND LOCATIONS:
Overall Officials: Laurence Hirsch, MD, Study Director — Becton Dickinson, World Wide VP Diabetes Care
Locations (4):
- United States (4):
  - AMCR Institute Inc., Escondido, California
  - Atlanta Diabetes Associates, Atlanta, Georgia
  - Rocky Mountain Diabetes and Osteoporosis Center, Idaho Falls, Idaho
  - TKL Research, Fair Lawn, New Jersey

IPD SHARING:
Plan to Share IPD: No